CLINICAL TRIAL: NCT03056417
Title: Impact of Lifestyle Changes Via the Complete Health Improvement Program on Telomerase Activity and Telomere Length in Patients With Chronic Pain
Brief Title: Impact of Lifestyle Changes on Telomeric Activity in Patients With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14X145
Record Dates: First submitted 2017-02-13; First posted 2017-02-17 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-09

CONDITIONS: Chronic Pain
Keywords: chronic pain; telomere; telomerase; life style
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the Complete Health Improvement Program.
  Interventions: Behavioral: The Complete Health Improvement Program
- No Change to Treatment (No Intervention): Participants who choose not to participate in the Complete Health Improvement Program.

INTERVENTIONS:
Behavioral: The Complete Health Improvement Program — The Complete Health Improvement Program is a nationally recognized program that encourages a diet of whole plant based foods, moderate exercise, stress reduction, and social support.
  Arms: Intervention

SUMMARY:
The current project will use the Complete Health Improvement Program (CHIP) as an intervention for patients with chronic pain. CHIP is a nationally recognized program that encourages a diet of whole plant-based foods, moderate exercise, stress reduction, and social support. Patients with chronic pain who enroll in CHIP classes will be monitored and compared to patients with chronic pain who are not enrolled in CHIP classes. It is hypothesized that patients who complete CHIP will have increased telomerase activity and longer relative telomere length at follow-up when compared to those who do not enroll in the program. Chromosomes consist of DNA that contains the genetic makeup of an individual; and telomeres are the caps on these chromosomes that protect them from damage. Telomere shortening occurs normally with aging and once they are too short to replicate cellular death occurs. Telomerase is a ribonucleic protein that counterbalances this shortening by extending the ends of chromosomes. Research has shown that patients with chronic pain may have shorter telomeres relative to others of the same age. This study will investigate this association further.

ELIGIBILITY:
Inclusion Criteria:

* 40-70 years old
* Physician confirmed chronic pain diagnosis for at least 6 months

Exclusion Criteria:

* Pregnancy
* Physical or mental condition that limits ability to provide consent or answer questionnaires

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Telomerase activity changes as a result of lifestyle change | Change from baseline telomerase at 3 months
  Assessed via peripheral blood mononuclear cells
Subjective pain ratings as a function of positive lifestyle modifications | Change from baseline subjective pain at 3 months
  Assessed via the Brief Pain Inventory - Short Form. Measures pain intensity from 0 to 10, 10 being pain as bad as you can imagine. Also measures the extent to which pain interferes with daily functioning (0 - 10 possible, with 10 indicating completely interferes).

SECONDARY OUTCOMES:
Relative telomere length changes as a result of lifestyle change | Change from baseline telomere length at 3 months
  Assessed via whole blood samples
Relative telomere length changes as a result of lifestyle change at 1-year follow-up | Change from 3 month follow-up data of telomere length at 1-year
  Assessed via whole blood samples
Fasting glucose changes as a result of lifestyle change | Change from baseline fasting glucose at 3 months
  Assessed via whole blood samples
Fasting glucose changes as a result of lifestyle change at 1-year follow-up | Change from 3 month follow-up data of fasting glucose at 1-year
  Assessed via whole blood samples
Fasting lipid profile (i.e., HDL, LDL, triglycerides) modification as a result of lifestyle change | change from baseline fasting lipids at 3 months
  Assessed via whole blood
Fasting lipid profile (i.e., HDL, LDL, triglycerides) modification as a result of lifestyle change at 1-year follow-up | Change from 3 month follow-up data of fasting lipids at 1-year
  Assessed via whole blood
C-reactive protein changes as a result of lifestyle change | change from baseline C-reactive protein at 3 months
  Assessed via plasma
C-reactive protein changes as a result of lifestyle change at 1-year follow-up | Change from 3 month follow-up data of C-reactive protein at 1-year
  Assessed via plasma
Overall well-being changes as a result of lifestyle change | change from baseline overall well-being at 3 months
  The RAND-36 item short form survey. High score indicates more favorable health state. Minimum score 0 Maximum score 100.
Overall well-being changes as a result of lifestyle change at 1-year follow-up | Change from 3 month follow-up data of overall well-being at 1-year
  The RAND-36 item short form survey. High score indicates more favorable health state. Minimum score 0 Maximum score 100.
Perceived Stress changes as a result of lifestyle change | change from baseline perceived stress at 3 months
  The 14-item Perceived Stress Scale. Minimum score 0 Maximum score 40. Higher scores indicate greater perceived stress.
Perceived Stress changes as a result of lifestyle change at 1-year follow-up | Change from 3 month follow-up data of perceived stress at 1-year
  The 14-item Perceived Stress Scale. Minimum score 0 Maximum score 40. Higher scores indicate greater perceived stress.
Depressive symptom changes as a result of lifestyle change | change from baseline depressed mood at 3 months
  Center for Epidemiological Studies Depression Scale. Higher score indicates greater depressed mood. Minimum score 0 Maximum score 60.
Depressive symptom changes as a result of lifestyle change at 1-year follow-up | Change from 3 month follow-up data of depressed mood at 1-year
  Center for Epidemiological Studies Depression Scale. Higher score indicates greater depressed mood. Minimum score 0 Maximum score 60.
Perceived social support modification as a result of lifestyle change | change from baseline perceived social support at 3 months
  Multidimensional Scale of Perceived Social Support. Higher score indicates greater perceived social support. Minimum score 1 Maximum score 7.
Perceived social support modification as a result of lifestyle change at 1-year follow-up | Change from 3 month follow-up data of perceived social support at 1-year
  Multidimensional Scale of Perceived Social Support. Higher score indicates greater perceived social support. Minimum score 1 Maximum score 7.
Health-Promoting behavior change as a result of lifestyle modification | change from baseline health promoting behavior at 3 months
  Health-Promoting Lifestyle Profile II questionnaire. Higher score indicate greater health promotion. Minimum score 1 Maximum score 4.
Health-Promoting behavior change as a result of lifestyle modification at 1-year follow-up | Change from 3 month follow-up data of health promoting behavior at 1-year
  Health-Promoting Lifestyle Profile II questionnaire. Higher score indicate greater health promotion. Minimum score 1 Maximum score 4.
Telomerase activity changes as a result of lifestyle change at 1-year follow-up | Change from 3 month follow-up data of telomerase activity at 1-year
  Assessed via peripheral blood mononuclear cells
Subjective pain ratings as a function of positive lifestyle modifications at 1-year follow-up | Change from 3 month follow-up data of subjective pain at 1-year
  Assessed via the Brief Pain Inventory - Short Form. Measures pain intensity from 0 to 10, 10 being pain as bad as you can imagine. Also measures the extent to which pain interferes with daily functioning (0 - 10 possible, with 10 indicating completely interferes).

CONTACTS AND LOCATIONS:
Overall Officials: Katrina Hamilton, M.S., Principal Investigator — Ohio University; David Drozek, D.O., Study Director — Ohio University; Peggy Zoccola, Ph.D., Study Chair — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shcherbakova DM, Zvereva ME, Shpanchenko OV, Dontsova OA. [Telomerase: structure and properties of the enzyme, characteristics of the yeast telomerase]. Mol Biol (Mosk). 2006 Jul-Aug;40(4):580-94. Russian. PMID 16913218
- [Background] Li B, Comai L. Requirements for the nucleolytic processing of DNA ends by the Werner syndrome protein-Ku70/80 complex. J Biol Chem. 2001 Mar 30;276(13):9896-902. doi: 10.1074/jbc.M008575200. Epub 2001 Jan 4. PMID 11152456
- [Background] Drozek D, Diehl H, Nakazawa M, Kostohryz T, Morton D, Shubrook JH. Short-term effectiveness of a lifestyle intervention program for reducing selected chronic disease risk factors in individuals living in rural appalachia: a pilot cohort study. Adv Prev Med. 2014;2014:798184. doi: 10.1155/2014/798184. Epub 2014 Jan 16. PMID 24527219
- [Background] Hassett AL, Epel E, Clauw DJ, Harris RE, Harte SE, Kairys A, Buyske S, Williams DA. Pain is associated with short leukocyte telomere length in women with fibromyalgia. J Pain. 2012 Oct;13(10):959-69. doi: 10.1016/j.jpain.2012.07.003. PMID 23031395